CLINICAL TRIAL: NCT01382381
Title: Evaluation of Implanted Aortic Arch and Branch Pulmonary Artery Stents Durability and Function
Brief Title: Intravascular Stents Fracture Effects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Avraham Lorber, Head, Pediatric Cardiology and Adults with Congenital Heart Disease, Rambam Medical Center, P.O.B 9602, Haifa 31096, Israel, Prof. Avraham Lorber, Head, Pediatric Cardiology and Adults with Congenital Heart Disease, Rambam Medical Center, P.O.B 9602, Haifa 31096, Israel
Other Study IDs: 0081CTIL
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-02

CONDITIONS: Durability of Implanted Intravascular Stents; Hemodynamic Effect of Implanted Intravascular Stents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to evaluate long term durability and hemodynamic effect of implanted stents in the aortic arch and in pulmonary artery branches.

DETAILED DESCRIPTION:
Patients who underwent trans-catheter implantation of balloon expanded stents in the aortic arch and in branch pulmonary arteries will be evaluated by physical examination with blood pressure values measurement of upper and lower limbs.

Echo-Doppler cardiography will be performed for flow velocity analysis. Zoomed fluoroscopy will be performed and recorded in two orthogonal views to evaluate stent integrity or stent fracture.

It is our intention to include 20 patients in this study from our follow-up clinic.

ELIGIBILITY:
Inclusion Criteria:

-patients who underwent stent implantation for coarctation of the aorta and for branch pulmonary artery stenosis

Exclusion Criteria:

-Pregnancy

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty patients who underwent stent implantation for coarctation of the aorta and for branch pulmonary artery stenosis will be recruited for the study from our out-patients follow-up clinic
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Study Completion 2012-07 (Estimated)